CLINICAL TRIAL: NCT06495619
Title: Effectiveness of Integrative Intervention Strategies for Binge Eating in Patients With Overweight or Obesity: A Multidisciplinary Approach
Brief Title: Integrative Intervention Strategies for Binge Eating in Patients With Overweight or Obesity
Acronym: BE-side
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, CHIARA CONTI, Associate professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prot. n. 254
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Binge Eating; Overweight and Obesity
Keywords: Binge Eating; Overweight; Obesity; Guided Self-Help; Biofeedback
MeSH Terms: conditions — Bulimia; Overweight; Obesity | interventions — Glutathione; Biofeedback, Psychology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (1)TAU (Active Comparator): treatment-as-usual for weight loss (TAU)
  Interventions: Behavioral: treatment-as-usual
- (2)TAU+GSH (Active Comparator): combined TAU and guided self-help for improving eating behaviors (TAU+GSH)
  Interventions: Behavioral: combined TAU and guided self-help
- (3)TAU+GSH+BF (Active Comparator): combined TAU, GSH, and biofeedback (TAU+GSH+BF)
  Interventions: Behavioral: combined TAU, GSH, and biofeedback

INTERVENTIONS:
Behavioral: treatment-as-usual — life style modification intervention for weight loss
  Other Names: TAU
  Arms: (1)TAU
Behavioral: combined TAU and guided self-help — combined TAU and guided self-help for improving eating behaviors
  Other Names: TAU+GSH
  Arms: (2)TAU+GSH
Behavioral: combined TAU, GSH, and biofeedback — combined TAU, GSH, and biofeedback for improving eating behaviors and interoceptive awareness and arousal regulation
  Other Names: TAU+GSH+BF
  Arms: (3)TAU+GSH+BF

SUMMARY:
The main goal of the clinical trial is to compare the short- and long-term outcomes of three 12-week interventions among outpatients with overweight/obesity and binge eating (BE):

1. treatment-as-usual for weight loss (TAU);
2. combined TAU and guided self-help for improving eating behaviors (TAU+GSH);
3. combined TAU, GSH, and biofeedback (TAU+GSH+BF). The primary outcomes will be self-reported reduction of days with objective BE episodes (OBEs).

The secondary outcomes will be impulsivity, emotion dysregulation, interoceptive awareness, distress, physiological correlates of arousal (skin conductance and heart rate variability), and inflammatory biomarkers.

The TAU+GSH arm is expected to be comparable to the TAU+GSH+BF arm in reducing the number of days with OBEs but is expected to be significantly less effective in improving secondary outcomes (impulsivity, emotional dysregulation, interoceptive awareness, distress, physiological inflammatory markers). The TAU arm is expected to show significant inferiority regarding the primary and secondary outcomes and cost-effectiveness compared to the TAU+GSH and TAU+GSH+BF conditions.

ELIGIBILITY:
Inclusion Criteria:(1) age 18-65 years; (2) BMI≥25 kg/m2; (3) ability to read and write in Italian; (4) Binge Eating Disorder (BED) or subthreshold BED status.

-

Exclusion Criteria: (1) current treatment for BE with a registered psychologist; (2) severe psychiatric disorders; (4) cognitive impairment; (5) pregnancy; (6) severe medical comorbidity.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
objective BE episodes (OBEs) | 12-week follow-up-1 4-month follow-up-2 (after the end-of-treatment)
  The primary outcomes will be self-reported reduction of days with objective BE episodes (OBEs)

SECONDARY OUTCOMES:
psychological variables | (T0) baseline; (T1)12-week follow-up-1; (T2) 4-month follow-up-2 (after the end-of-treatment)
  The secondary outcomes will be impulsivity, emotion dysregulation, interoceptive awareness, distress.
physiological correlates of arousal | (T0) baseline; (T1)12-week follow-up-1; (T2) 4-month follow-up-2 (after the end-of-treatment)
  The secondary outcomes will be skin conductance and heart rate variability.
inflammatory biomarkers | (T0) baseline; (T1)12-week follow-up-1; (T2) 4-month follow-up-2 (after the end-of-treatment)
  The secondary outcomes will be ClpB protein and IgG

IPD SHARING:
Plan to Share IPD: No
The data sets generated during and/or analysed during the current study are available from the PI on reasonable request.

REFERENCES:
- [Background] de Zwaan M, Herpertz S, Zipfel S, Tuschen-Caffier B, Friederich HC, Schmidt F, Gefeller O, Mayr A, Lam T, Schade-Brittinger C, Hilbert A. INTERBED: internet-based guided self-help for overweight and obese patients with full or subsyndromal binge eating disorder. A multicenter randomized controlled trial. Trials. 2012 Nov 21;13:220. doi: 10.1186/1745-6215-13-220. PMID 23171536
- [Background] DiMarco ID, Klein DA, Clark VL, Wilson GT. The use of motivational interviewing techniques to enhance the efficacy of guided self-help behavioral weight loss treatment. Eat Behav. 2009 Apr;10(2):134-6. doi: 10.1016/j.eatbeh.2009.02.001. Epub 2009 Feb 15. PMID 19447358
- [Background] Mueller J, Richards R, Jones RA, Whittle F, Woolston J, Stubbings M, Sharp SJ, Griffin SJ, Bostock J, Hughes CA, Hill AJ, Boothby CE, Ahern AL. Supporting Weight Management during COVID-19 (SWiM-C): twelve-month follow-up of a randomised controlled trial of a web-based, ACT-based, guided self-help intervention. Int J Obes (Lond). 2023 Jan;47(1):51-59. doi: 10.1038/s41366-022-01232-x. Epub 2022 Nov 11. PMID 36369513
- [Background] Varela C, Oda-Montecinos C, Andres A, Saldana C. Effectiveness of web-based feedback interventions for people with overweight and obesity: systematic review and network meta-analysis of randomized controlled trials. J Eat Disord. 2021 Jun 26;9(1):75. doi: 10.1186/s40337-021-00432-6. PMID 34174949
- [Background] de Zwaan M, Herpertz S, Zipfel S, Svaldi J, Friederich HC, Schmidt F, Mayr A, Lam T, Schade-Brittinger C, Hilbert A. Effect of Internet-Based Guided Self-help vs Individual Face-to-Face Treatment on Full or Subsyndromal Binge Eating Disorder in Overweight or Obese Patients: The INTERBED Randomized Clinical Trial. JAMA Psychiatry. 2017 Oct 1;74(10):987-995. doi: 10.1001/jamapsychiatry.2017.2150. PMID 28768334
- [Background] Frank DL, Khorshid L, Kiffer JF, Moravec CS, McKee MG. Biofeedback in medicine: who, when, why and how? Ment Health Fam Med. 2010 Jun;7(2):85-91. PMID 22477926